CLINICAL TRIAL: NCT00831714
Title: Xarelto in the Prophylaxis of Post Surgical Venous Thromboembolism After Elective Major Orthopedic Surgery of Hip or Knee
Brief Title: Xarelto for VTE Prophylaxis After Hip or Knee Arthroplasty
Acronym: XAMOS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13802; XA0801 (Other: company internal)
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thromboembolism
Keywords: Prophylaxis of Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Group 2
  Interventions: Drug: Standard care treatment for VTE prophylaxis

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Female and male patients, who are at least 18 years of age and will undergo elective hip or knee arthroplasty, after the decision for VTE prophylaxis with Rivaroxaban has been made
  Groups: Group 1
Drug: Standard care treatment for VTE prophylaxis — Female and male patients, who are at least 18 years of age and will undergo elective hip or knee arthroplasty, after the decision for a pharmacologic VTE prophylaxis treatment other than rivaroxaban has been made
  Groups: Group 2

SUMMARY:
The main goal is to provide additional information to the risk-benefit assessment of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who will undergo elective hip or knee arthroplasty.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients, who are at least 18 years of age and will undergo elective hip or knee arthroplasty, after the decision for a pharmacologic VTE prophylaxis treatment has been made
Sampling Method: Probability Sample
Enrollment: 19076 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Data collection on: Bleeding events reported as serious or non-serious adverse events; Symptomatic thromboembolic events (DVT, PE) reported as adverse events; Uncommon adverse events (incidence rate between 0.1 % and 1 %); All cause mortality | During observation period of three months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (42):
- Many Locations, Australia
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Bosnia and Herzegovina
- Many Locations, Brazil
- Many Locations, Canada
- Many Locations, Chile
- Many Locations, China
- Many Locations, Colombia
- Many Locations, Cyprus
- Many Locations, Czechia
- Many Locations, Denmark
- Many Locations, Estonia
- Many Locations, Finland
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Hong Kong
- Many Locations, Hungary
- Many Locations, India
- Many Locations, Italy
- Many Locations, Latvia
- Many Locations, Lebanon
- Many Locations, Lithuania
- Many Locations, Mexico
- Many Locations, Netherlands
- Many Locations, North Macedonia
- Many Locations, Norway
- Many Locations, Philippines
- Many Locations, Portugal
- Many Locations, Serbia
- Many Locations, Singapore
- Many Locations, Slovakia
- Many Locations, South Africa
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Switzerland
- Many Locations, United Arab Emirates
- Many Locations, United Kingdom
- Many Locations, Venezuela
- Many Locations, Vietnam

REFERENCES:
- [Background] Turpie AG, Haas S, Kreutz R, Mantovani LG, Pattanayak CW, Holberg G, Jamal W, Schmidt A, van Eickels M, Lassen MR. A non-interventional comparison of rivaroxaban with standard of care for thromboprophylaxis after major orthopaedic surgery in 17,701 patients with propensity score adjustment. Thromb Haemost. 2014 Jan;111(1):94-102. doi: 10.1160/TH13-08-0666. Epub 2013 Oct 24. PMID 24154549
- [Derived] Turpie AG, Schmidt AC, Kreutz R, Lassen MR, Jamal W, Mantovani L, Haas S. Rationale and design of XAMOS: noninterventional study of rivaroxaban for prophylaxis of venous thromboembolism after major hip and knee surgery. Vasc Health Risk Manag. 2012;8:363-70. doi: 10.2147/VHRM.S30064. Epub 2012 Jun 1. PMID 22701330